CLINICAL TRIAL: NCT04087993
Title: Randomised, Open Lable, Active Controlled Clinical Trial to Demonstrate Safety and Efficacy of an i.v. Administration of Polyglucoferron Compared to i.v. Ferric Carboxymaltose and Oral Iron Substitution in Preoperative Treatment of Iron Deficiency Anaemia in Patients With Elective Non-cardiac Surgery (IDA I)
Brief Title: Polyglucoferron Compared to i.v. Ferric Carboxymaltose and Oral Iron Substitution in Preoperative Treatment of Iron Deficiency Anaemia in Patients
Acronym: IDA-I
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: difficult recruitment - redesign in discussion
Sponsor: Dr. Frank Behrens (Other)
Collaborators: University Hospital Frankfurt, Department of Anaesthesiology (Unknown); IRON4U (Unknown); University Hospital Frankfurt Institute for Biostatistics & Mathematical Modelling (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Sponsor representative, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP0916_02
Record Dates: First submitted 2019-08-29; First posted 2019-09-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Iron Deficiency Anemia
Keywords: pre surgery iron treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: 2:2:1 distribution Polyglucoferron, Ferric Carboxymaltose i.v., or oral iron substitution with Ferrous sulfate. After safety assessment of first 35 patients treated with Polyglucoferron or Ferric Carboxymaltose i.v. respectively, Ferric Carboxymaltose arm will be closed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polyglucoferron (Experimental): once intravenously, dosing according to Hb-levels and body weight, 500 - 2000 mg
  Interventions: Drug: Polyglucoferron
- Ferric Carboxymaltose (Active Comparator): Once intravenously (a second administration is allowed), dosing according to Hb-levels and body weight (500 - 2000 mg, max. single dose of 1000 mg)
  Interventions: Drug: Ferric carboxymaltose
- Ferrous sulfate (Active Comparator): capsules, orally, dosing 50 mg - 200 mg (50 mg: 1 capsule in total, 200 mg: 4 capsules in total, taken as 2 capsules twice daily), duration of treatment 28 days
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Polyglucoferron — intravenous administration
  Other Names: Feramyl
  Arms: Polyglucoferron
Drug: Ferric carboxymaltose — intravenous administration
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose
Drug: Ferrous Sulfate — oral administration
  Other Names: Ferro sanol duodenal
  Arms: Ferrous sulfate

SUMMARY:
Patients with IDA and for whom fast replenishment of iron stores is necessary, e.g. if its not appropriated to postpone surgery, will be identified within 28 to 42 days before surgery. Patients will be randomised to receive either Polyglucoferron intravenously (i.v.), Ferric Carboxymaltose i.v. or oral iron substitution with Ferrous sulfate.

DETAILED DESCRIPTION:
Randomised, active-controlled, open-labelled, parallel group, multicentre study to demonstrate superiority of Polyglucoferron i.v. compared to oral iron substitution for the treatment of iron deficient anaemic patients who need fast replenishment of iron stores as judged by the treating physician, e.g. if it is not appropriate to postpone surgery, before elective non-cardiac surgery and superiority of Polyglucoferron i.v. vs Ferric Carboxymaltose in short term safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; aged ≥ 18 years
* Planned to undergo non-cardiac surgery (e.g., orthopaedic, vascular, visceral surgery) within 28 to 42 days, which requires a fast replenishment of the patients' iron stores (e.g.if it is not appropriate to postpone surgery) as judged by the treating physician
* Iron deficiency defined as s-ferritin <100 ng/mL and s-transferrin saturation <20%
* Relevant anaemia defined as haemoglobin of <12 g/dL for female and <13 g/dL for men
* Written informed consent; willing and able to comply with the protocol

Exclusion Criteria:

* Pregnancy in female patients or breastfeeding women
* Female patients not willing to use a safe method of contraception (PEARL index <1) for the full study period
* Severe anaemia with Hb < 8 g/dL
* Any ingoing bleeding as judged by the treating physician
* Patients receiving blood transfusion 24 weeks prior screening
* Severe physical inability, e.g., American Society of Anesthesiologists (ASA) physical status IV or V
* Haematuria and proteinuria of unknown or known origin
* Non-iron deficiency anaemia, e.g., known Vitamin B12 or folate deficiency, haemoglobinopathy, or unexplained anaemia
* Anticipated medical need for erythropoiesis-stimulating agents during the study period
* Patients with any contraindication to the investigational products, e.g.,

  1. known sensitivity to iron or an ingredient of the investigational products
  2. History of systemic allergic reactions
  3. Haemachromatosis, thalassemia or TSAT >50% as indicator of iron overload
  4. Acute or chronic intoxication
  5. Infection (patient on non-prophylactic antibiotics)
  6. Chronic liver disease and/or screening Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) above three times the upper limit of the normal range
* Chronic kidney disease, defined as Glomerular Filtration Rate (GFR) <30 mL/min
* Serum Creatinine > 150 μmol/L
* Active uncontrolled immune-mediated diseases such as rheumatoid arthritis or inflammatory bowel disease
* Primary haematologic disease
* Drug or alcohol abuse according to WHO definition
* Potentially unreliable patients, and those judged by the investigator to be unsuitable for the study
* Current or previous participation in another clinical trial during the last 90 days before screening
* Exclusion criteria related to Ferrous sulfate

  1. according to summary of product characteristics (SmPC)
  2. hypersensitivity to any ingredient in the formulation
  3. concomitant parenteral iron
  4. haemochromatosis, and other iron overload syndromes
* Exclusion criteria related to Ferric Carboxymaltose:

  1. according to SmPC
  2. hypersensitivity to the active substance, to Ferinject or any of its excipients
  3. known serious hypersensitivity to other parenteral iron products
  4. anaemia not attributed to iron deficiency
  5. evidence of iron overload or disturbances in the utilisation of iron
* Exclusion criteria related to Polyglucoferron f) hypersensitivity to any ingredient in the formulation

  1. known serious hypersensitivity to other parenteral iron products
  2. anaemia not attributed to iron deficiency
  3. evidence of iron overload or disturbances in the utilisation of iron

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Normalisation or Increase of hemaglobin(Hb)-level | baseline (BL) to day before surgery (visit 4)
  Proportion of patients achieving normalized Hb-levels (according to World Health Organization (WHO) definition) or an increase of at least 1.5 g/dl Hb at day before surgery (visit 4) compared to baseline (BL) in the Polyglucoferron treatment arm compared to oral iron substitution with Ferrous sulfate
Detection of urine iron | approx. 8 hours
  Detection of urine iron in the first urine after the end of i.v. administration, defined as short term safety surrogate marker after administration of the i.v. treatments

SECONDARY OUTCOMES:
Units of allogenic red blood cell transfusion | baseline to visit 5 approx. 70 day
  Proportion of units of allogenic red blood cell transfusion from BL until visit 5
Hb values | baseline to visit 4 approx. 35 day
  Mean change in Hb at visit 4 compared to BL
Hb values | baseline to visit 5 approx. 70 day
  Mean change in Hb at visit 5 compared to BL
Transferrin Saturation (TSAT) values | baseline to visit 5 approx. 70 day
  Mean change in TSAT at visit 5 compared to BL
Transferrin Saturation (TSAT) values | baseline to visit 4 approx. 35 day
  Mean change in TSAT at visit 4 compared to BL
iron values | baseline to visit 4 approx. 35 day
  Mean change in serum iron at visit 4 compared to BL
iron values | baseline to visit 5 approx. 70 day
  Mean change in serum iron at visit 5 compared to BL
ferritin values | baseline to visit 5 approx. 70 day
  Mean change in serum ferritin at visit 5 compared to BL
ferritin values | baseline to visit 4 approx. 35 day
  Mean change in serum ferritin at visit 4 compared to BL
transferrin values | baseline to visit 4 approx. 35 day
  Mean change in serum ferritin at visit 4 compared to BL
transferrin values | baseline to visit 5 approx. 70 day
  Mean change in serum ferritin at visit 5 compared to BL
number of adverse events (AE)/serious adverse events (SAE) | baseline to 28 days after surgery, approx. 56 days
  Tolerability measured by overall number of AEs/SAEs until 28 days after surgery
incidence of adverse events (AE)/serious adverse events (SAE) | baseline to 28 days after surgery, approx. 56 days
  Tolerability by incidence of AEs/SAEs until 28 days after surgery
Seriousness of adverse events (AE)/serious adverse events (SAE) | baseline to 28 days after surgery, approx. 56 days
  Overall tolerability by seriousness of AEs/SAEs until 28 days after surgery
Relationship of adverse events (AE)/serious adverse events (SAE) | baseline to 28 days after surgery, approx. 56 days
  Overall tolerability by relationship of AEs/SAEs until 28 days after surgery
Severity of adverse events (AE)/serious adverse events (SAE) | baseline to 28 days after surgery, approx. 56 days
  Overall tolerability by severity of AEs/SAEs until 28 days after surgery
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes White blood count on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in thrombocytes on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in serum creatinine on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in AST on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in ALT on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in gamma GT on each visit
Changes in Laboratory parameters | throughout study conduction, max 77 days
  Changes in phosphate on each visit
Changes in vital signs | throughout study conduction, max 77 days
  Changes in vital signs on each visit
Changes in blood pressure | throughout study conduction, max 77 days
  Changes in blood pressure on each visit
Changes in heart rate | throughout study conduction, max 77 days
  Changes in heart rate on each visit
Changes in physical exam | throughout study conduction, max 77 days
  Changes in physical exam on each visit
adverse events related to administration | at baseline
  AEs related to injection/infusion site reactions (i.v. group only)
adverse events related to administration | 7 days after baseline, at Visit 3
  AEs related to injection/infusion site reactions (i.v. group only)
hypersensitivity reactions | at baseline
  documentation of anaphylatic or anaphylactoid reactions (i.v. group only)
hypersensitivity reactions | at study visit 3
  documentation of anaphylatic or anaphylactoid reactions (i.v. group only)
Mortality | within 28 days after surgery, approx. 56 days
  All-cause mortality within 28 days after surgery
Quality of Life (SF36) | base line to visit 4 approx 35 days
  Assessment of Quality of Life by SF36 questionnaire at visits 4 compared to BL
Quality of Life (SF36) | baseline to visit 5 approx 70 days
  Assessment of Quality of Life by SF36 questionnaire at visits 5 compared to BL
Duration of hospital stay | 28 days
  Duration of hospital stay (days) until 28 days after surgery
Number of patients with normalized Hb-values | baseline to visit 4 approx 35 days
  Number of patients with normalized Hb-values after iron substitution (n, %) at visits 4 and 5
Number of patients with normalized Hb-values | baseline to visit 5 approx 70 days
  Number of patients with normalized Hb-values after iron substitution (n, %) at and 5
Analysis of total iron levels | approx 4 hours
  Analysis of total iron levels in plasma at BL after end of iron administration (for the i.v. groups (safety analysis group) only)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, Prof. MD, Principal Investigator — University Hospital of Goethe-University Frankfurt
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital of Goethe-University, Frankfurt, Hessia, Germany